CLINICAL TRIAL: NCT05731765
Title: Automated Detection of Spontaneous Venous Pulsations Within Fundal Videos Using Machine Learning
Brief Title: SVP Detection Using Machine Learning
Acronym: SVP-ML
Status: Active, not recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2023-01-30; First posted 2023-02-16 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Intracranial Pressure Increase
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients aged ≥18 years with presumed normal intracranial pressure
  Interventions: Diagnostic Test: Machine Learning Model
- Patients aged ≥18 years with suspected raised intracranial pressure
  Interventions: Diagnostic Test: Machine Learning Model

INTERVENTIONS:
Diagnostic Test: Machine Learning Model — Automated machine learning system for the detection of spontaneous venous pulsations and quantification of intracranial pressure

SUMMARY:
This diagnostic study will use 410 retrospectively captured fundal videos to develop ML systems that detect SVPs and quantify ICP. The ground truth will be generated from the annotations of two independent, masked clinicians, with arbitration by an ophthalmology consultant in cases of disagreement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with presumed normal ICP undergoing routine dilated OCT scans.
* Patients undergoing a LP or continuous ICP monitoring with implanted transcranial pressure transducer devices at in- or out-patient neurology, neurosurgery or neuro-ophthalmology services.

Exclusion Criteria:

* Glaucoma diagnosis or glaucoma suspects in either eye.
* Bilateral restricted fundal view, e.g. advanced bilateral cataracts.
* Bilateral retinal vein or artery occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with presumed normal ICP or suspected raised ICP
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Area-under-the receiver operating characteristic (AUROC) for spontaneous venous pulsations detection | 1 year
  Binary classification performance of the machine learning model

SECONDARY OUTCOMES:
Localisation of spontaneous venous pulsations | 1 year
  Bounding box overlap for the machine learning model
Quantification of intracranial pressure | 1 year
  Mean absolute error for the prediction of the intracranial pressure

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data would be shared, where possible, through a restricted-access data sharing agreement, where in line with KCL data governance requirements.
Supporting Information: Study Protocol
Time Frame: Within 12 months of study completion
Access Criteria: Data sharing agreement and data governance